CLINICAL TRIAL: NCT05535777
Title: Improving Influenza Vaccination Delivery Across a Health System by the Electronic Health Records Patient Portal RCT 5 (LADHS)
Brief Title: Patient Portal Flu Vaccine Reminders_RCT 5 (LADHS)
Acronym: LADHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Los Angeles County Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Executive Vice Chair, Vice Chair for Research, UCLA David Geffen School of Medicine, Department of Pediatrics, University of California, Los Angeles, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-001889-00016 (LADHS); R01AI135029 (NIH)
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Influenza; Respiratory Tract Infections
Keywords: Reminder Recall (R/R); Influenza Vaccine; Electronic Health Record; Text Message; Vaccine
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Pragmatic comparative effectiveness trial with a standard-of-care control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Text Reminders with Callback by Person (Active Comparator): Participants in this arm will receive up to 3 R/R messages by text. R/R message will receive a phone call back by a call center agent if they press "1" in response to a question on the original text message. The call center agent's job is to schedule patients for clinical visits. These call center agents will be trained by our faculty and staff and will have the usual HIPAA and other patient confidentiality training.
  Interventions: Behavioral: Enhanced texts with Callback by a Person
- Enhanced Bidirectional Text Reminders (Active Comparator): Participants in this arm will receive a text message from a call center agent if they press "1" in response to a question on the original text message. The bidirectional texts will have an agent who can answer questions and schedule an appointment through text message back-and-forth conversations with the patient. Bidirectional texts will be exchanged on a HIPAA compliant bidirectional text messaging platform. The patient will use the regular SMS function on their cellphone and the agent will receive and respond to the bidirectional text on the HIPAA compliant platform.
  Interventions: Behavioral: Enhanced Bidirectional Texts
- Standard Text Reminders (No Intervention): Participants in this arm will receive up to 3 text messages, reminding them about the importance of influenza vaccination. The standard texts will include a clinic call back number and patient portal self-scheduling for patients to schedule their influenza vaccines. The direct scheduling texts includes a direct number to an agent that can help schedule and answer questions on the phone in real time. The texts with a direct number to schedule will link a specified phone number to call and schedule. This number would be answered by a central agent quickly and a patient could schedule their flu shot at any clinic site. This specific phone number would not go through the multiple option menus a patient would normally experience when calling their clinic.

INTERVENTIONS:
Behavioral: Enhanced texts with Callback by a Person — Enhanced texts - Callback by a person: Patient randomized to this study arm will receive a phone call back by a call center agent if they press "1" in response to a question on the original text message. The call center agent's job is to schedule patients for clinical visits. These call center agents will be trained by our faculty and staff and will have the usual HIPAA and other patient confidentiality training.
  Arms: Enhanced Text Reminders with Callback by Person
Behavioral: Enhanced Bidirectional Texts — Patients randomized to this study arm will receive a text message from a call center agent if they press "1" in response to a question on the original text message. The bidirectional texts will have an agent who can answer questions and schedule an appointment through text message back-and-forth conversations with the patient.
  Arms: Enhanced Bidirectional Text Reminders

SUMMARY:
This trial is taking place in Los Angeles, CA at clinics within the Los Angeles Department of Health clinics.

The study design is a comparative effectiveness trial design. Patients will be randomized into 1) receiving enhanced texting with a callback by a trained call-center staff member to schedule a vaccine visit if the patient presses "1" in response to the text, 2) receiving enhanced bidirectional texting with a texting response from a trained call-center staff member who will help the patient schedule a vaccine visit through a series of back-and-forth texts, or 3) standard text reminders (control group). Patients in all arms will receive reminders if they are due for influenza vaccine.

Despite the Advisory Committee on Immunization Practices (ACIP) recommendation in 2010 that all people above 6 months of age should receive an annual flu vaccine, vaccination rates remain low: at 6m-4.9 yrs. (70%), 5-17.9 yrs. (56%), 18-64.9 yrs. (38%), and >65 yrs. (63%). The investigators will assess the effectiveness of enhanced text R/R messages as compared to the standard of care control (standard text reminders).

DETAILED DESCRIPTION:
Sub-optimal vaccination rates are a significant problem in the U.S., despite their effectiveness in preventing morbidity and mortality from vaccine-preventable illness. For influenza specifically, annual epidemics of influenza cause substantial morbidity in the U.S. with up to 40,00-80,000 deaths/year and many hospitalizations, emergency and outpatient visits, and significant costs.

Reminder/recall (R/R), sent by phone, mail or other modality, can improve child and adult influenza vaccination rates. However, the majority of pediatric or adult primary care practices do not conduct R/R. Barriers are lack of finances, personnel, and algorithms to identify eligible patients.

A technological breakthrough that might overcome these barriers involves patient text messaging at the health system level.

This randomized controlled trial will assess the effectiveness of reminders messages sent by text encouraging influenza vaccination, on increasing influenza vaccination rates within a health system. Patients will be randomized into three groups: 1) one-third of patients will receive enhanced text reminder messages, 2) one-third will receive enhanced bidirectional text reminder messages and 3) one-third will received standard-of-care text reminder messages.

Enhanced texts - Callback by a person: Patient randomized to this study arm will receive a phone call back by a call center agent if they press "1" in response to a question on the original text message. The call center agent's job is to schedule patients for clinical visits. These call center agents will be trained by our faculty and staff and will have the usual HIPAA and other patient confidentiality training.

Enhanced Bidirectional Texts: These texts are designed to help schedule a vaccine visit. Patients randomized to this study arm will receive a text message from a call center agent if they press "1" in response to a question on the original text message. The bidirectional texts will have an agent who can answer questions and schedule an appointment through text message back-and-forth conversations with the patient. Bidirectional texts will be exchanged on a HIPAA compliant bidirectional text messaging platform. The patient will use the regular SMS function on their cellphone and the agent will receive and respond to the bidirectional text on the HIPAA compliant platform.

Previous studies have shown that low-cost, behavioral nudges through texting can increase influenza vaccination uptake compared to usual care. However, there are limited studies that evaluate the effect of decreasing friction/barriers to scheduling especially within safety net populations. This study will examine the effect of strategies to reduce friction/barriers to scheduling including bidirectional text messages, and texts for patients to call for direct scheduling without wait time on influenza vaccination rates in adults within the 2022-2023 flu season.

For the primary analysis, the primary outcome will be the patient's end of flu season vaccination status. Intervention effects will be assessed using multivariable log-binomial regression models. Regressions will include indicators for each intervention as fixed effects, with the standard text condition as the reference group, and potentially clinic random effects, depending on retrospective analysis results. Models will also adjust for patient age, gender, race/ethnicity, insurance, and whether the patient was vaccinated in at least one of the prior two flu seasons.

The enhanced texts with callback, enhanced bidirectional texts, and standard-of-care text reminder messages will begin in September of 2022.

ELIGIBILITY:
Inclusion Criteria:

* LADHS patients identified as primary care patients assigned as follows: (1) assigned through managed care plans, (2) self-pay but linked with a provider, or (3) uninsured but assigned.

Exclusion Criteria:

* LADHS patient not identified as a primary care patient.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246295 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagyi, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Los Angeles County Department of Health Services, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enhanced Text Reminders With Callback by Person | Enhanced Bidirectional Text Reminders | Standard Text Reminders
Started | 6914 | 6901 | 180423
Completed | 6914 | 6901 | 180423
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Text Reminders With Callback by Person | Enhanced Bidirectional Text Reminders | Standard Text Reminders | Total
Number analyzed (Participants) | 6914 | 6901 | 180423 | 194238
Age, Customized [Count of Participants; unit: Participants]
  6 months+ | 6914 | 6901 | 180423 | 194238
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 3763 | 3638 | 96646 | 104047
  Male | 2927 | 3020 | 77372 | 83319
  Gender unspecified | 1 | 1 | 46 | 48
  Gender unknown | 3 | 1 | 36 | 40
  Missing | 220 | 241 | 6323 | 6784
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 8 | 216 | 232
  Asian | 415 | 383 | 9773 | 10571
  Black or African American | 764 | 729 | 19092 | 20585
  Hispanic/Latino | 4089 | 4135 | 108204 | 116428
  Multi-Race | 45 | 37 | 1166 | 1248
  Native Hawaiian or Other Pacific Islander | 15 | 9 | 279 | 303
  Other/Unknown | 1066 | 1061 | 27213 | 29340
  White | 292 | 298 | 8157 | 8747
  Missing | 220 | 241 | 6323 | 6784
Primary Language [Count of Participants; unit: Participants]
  English | 3656 | 3588 | 94207 | 101451
  Spanish | 2743 | 2759 | 71921 | 77423
  Other | 214 | 231 | 5669 | 6114
  Missing | 301 | 323 | 8626 | 9250
Vaccination in Prior Season [Count of Participants; unit: Participants]
  True | 1236 | 1272 | 33048 | 35556
  False | 5678 | 5629 | 147375 | 158682

OUTCOME MEASURES:

1. Primary Outcome: Receipt of the Annual Influenza Vaccine Among Adult and Pediatric Index Patients
Description: Percent of patients with annual influenza vaccination (between 9/1/22 - 4/1/23) among adult and pediatric index patients. Outcomes will be assessed via vaccine data extraction from the electronic health record and external claims and pharmacy data.
  The index patients must be an LADHS patient. Primary care patients who are empaneled to a primary care provider within DHS are assigned as follows: (1) assigned through managed care plans, (2) self-pay but linked with a provider or (3) uninsured but assigned). Individuals not affiliated with any primary care practice will be excluded from the primary analysis.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Text Reminders With Callback by Person | Enhanced Bidirectional Text Reminders | Standard Text Reminders
Number analyzed (Participants) | 6914 | 6901 | 180423
Participants | 4641 | 4629 | 120137

2. Secondary Outcome: Receipt of the Annual Influenza Vaccine Among Pediatric Index Patients
Description: Percent of patients with annual influenza vaccination (between 9/1/22 - 4/1/23) among pediatric index patients. Outcomes will be assessed via vaccine data extraction from the electronic health record and external claims and pharmacy data.
  The index patients must be an LADHS patient. Primary care patients who are empaneled to a primary care provider within DHS are assigned as follows: (1) assigned through managed care plans, (2) self-pay but linked with a provider or (3) uninsured but assigned). Individuals not affiliated with any primary care practice will be excluded from the primary analysis.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: We did not collect information regarding adverse events.
Description: We did not collect adverse event information. We monitored whether reminder recall through the portal and text was effective at increased influenza vaccination rates. Because influenza vaccination is recommended by the Advisory Committee on Immunization Practices and is part of the U.S. recommended vaccine schedule, we did not collect adverse event data.
Arm/Group | Enhanced Text Reminders With Callback by Person | Enhanced Bidirectional Text Reminders | Standard Text Reminders
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT05535777/Prot_SAP_000.pdf